CLINICAL TRIAL: NCT02028689
Title: A Phase 1, Randomized, Open-Label, Single-Dose Study to Evaluate Potential Pharmacokinetic Interaction Between Lesinurad and Metformin and Between Lesinurad and Furosemide in Health Adult Male Subjects
Brief Title: Metformin and Furosemide Drug-Drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RDEA594-128
Record Dates: First submitted 2013-10-17; First posted 2014-01-07 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
MeSH Terms: interventions — lesinurad; Metformin; Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lesinurad and Metformin (Experimental): Sequence A- Day 1: Metformin 850 mg; Day 5: Lesinurad 400 mg with metformin 850 mg
  Sequence B- Day 1: Lesinurad 400 mg with metformin 850 mg; Day 5: Metformin 850 mg
  Interventions: Drug: Lesinurad 400 mg; Drug: Metformin 850 mg
- Lesinurad and Furosemide (Experimental): Sequence C - Day 1: Furosemide 40 mg; Day 5: Lesinurad 400 mg with furosemide 40 mg
  Sequence D - Day 1: Lesinurad 400 mg with furosemide 40 mg; Day 5: Furosemide 40 mg
  Interventions: Drug: Lesinurad 400 mg; Drug: Furosemide 40 mg

INTERVENTIONS:
Drug: Lesinurad 400 mg
Drug: Metformin 850 mg
  Arms: Lesinurad and Metformin
Drug: Furosemide 40 mg
  Arms: Lesinurad and Furosemide

SUMMARY:
This study will assess the potential effects of lesinurad on the pharmacokinetics (PK) of metformin and furosemide in healthy, adult male subjects.

DETAILED DESCRIPTION:
Leinurad is a weak in vitro inhibitor of the hepatic transporter OCT1 and the renal transporters OAT1 and OAT3 (OAT1/3). To assess the clinical relevance of these in vitro findings, this clinical study will evaluate the effect of lesinurad on the PK of metformin (OCT1 substrate) and furosemide (OAT1/3 substrate).

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body weight ≥ 50 kg (110 lbs) and body mass index ≥ 18 and ≤ 30 kg/m2.
* Subject is free of any clinically significant disease or medical condition, per the Investigator's judgment.

Exclusion Criteria:

* Subject has a history or suspicion of kidney stones, prostatic hyperplasia, or urinary stricture.
* Subject has undergone major surgery within 3 months prior to Screening.
* Subject donated blood or experienced significant blood loss (>450 mL) within 12 weeks prior to Screening or gave a plasma donation within 4 weeks prior to Screening.
* Subject has inadequate venous access or unsuitable veins for repeated venipuncture.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
PK profile of metformin and furosemide from plasma | Day 1 and Day 5
  Profile in terms of maximum observed concentration (Cmax), time of occurence of maximum observed concentration (Tmax), area under the concentration-time curve (AUC), and apparent terminal half-life (t1/2).
PK profile of furosemide from urine | Day 1 and Day 5
  Profile in terms of renal clearance (CLr) and amount of compound excreted into urine unchanged (Ae).

SECONDARY OUTCOMES:
Incidence of Adverse Events and Changes in Laboratory, Electrocardiogram, and Vital Signs Parameters | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: S. Bradley, Study Director — Ardea Biosciences, Inc.
Locations (1):
- Kalamazoo, Michigan, United States